CLINICAL TRIAL: NCT06400264
Title: MATCH Treatment Subprotocol Z1M: Phase 2 Study of Nivolumab and BMS-986016 (Relatlimab) in Patients With LAG-3+ Tumors With Mismatch Repair Deficiency (MMR-d) After Progression on Anti-PD-1/PD-L1 Therapy
Brief Title: Testing Nivolumab and BMS-986016 (Relatlimab) as Potentially Targeting Treatment in Cancers That Are LAG-3+ and Have Mismatch Repair Deficiency (MATCH - Subprotocol Z1M)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No result will be reported- no patient accrued. Status Withdrawn: Study halted prematurely, prior to enrollment of first participant."
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01195; NCI-2024-01195 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1M (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1M (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-05-03; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Nivolumab; relatlimab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nivolumab and BMS-986016 [relatlimab]) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and BMS-986016 (relatlimab) over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients also undergo ECHO during screening as clinically indicated. Patients undergo a biopsy during screening and blood sample collection during screening and on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Biological: Relatlimab

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Biological: Relatlimab — Given IV
  Other Names: BMS-986016; BMS986016; Immunoglobulin G4, Anti-(human Lymphocyte Activation Gene-3 Protein) (Human Heavy Chain), Disulfide with Human Light Chain, Dimer

SUMMARY:
This phase II MATCH treatment trial tests how well nivolumab and BMS-986016 (relatlimab) works in treating patients with cancer that has certain genetic changes called LAG-3 mutations with mismatch repair deficiency. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as nivolumab and BMS-986016 (relatlimab), may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and BMS-986016 (relatlimab) over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and on study, as well as during follow-up as clinically necessary. Patients also undergo echocardiography (ECHO) during screening as clinically indicated. Patients undergo a biopsy during screening and blood sample collection during screening and on study.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must fulfill all eligibility criteria of MATCH Master Protocol at the time of registration to treatment step (Step 1, 3, 5, 7)
* Patients must have mismatch repair deficiency based on one of the following:

  * Mismatch repair testing done in any laboratory under Clinical Laboratory Improvement Act (CLIA) conditions with immunohistochemistry (IHC) for MLH1/MSH2 +/-MSH6 +/-PMS2 OR
  * Polymerase chain reaction (PCR)-based microsatellite testing using a validated assay done in any laboratory under CLIA conditions OR
  * A MATCH designated laboratory determination of mismatch repair (MMR) status by deoxyribonucleic acid (DNA) sequencing
* Patients must have LAG-3 expression at >= 1% as determined via the MATCH Master Protocol

  * NOTE: For patients entering the study, all patients must have LAG-3 testing performed as described in the MATCH Master Protocol. This includes patients entering the study via the outside assay process
* Patients with active melanoma are ineligible
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients must have Troponin T (TnT) or I (TnI) < 2 x upper limit of normal (ULN). Patients with TnT or TnI levels between > 1 to 2 x ULN will be allowed to register if repeat levels within 24 hours are =< 1 x ULN. If TnT or TnI levels are > 1 to 2 x ULN within 24 hours, the patients may undergo a cardiac evaluation and be considered for treatment. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 x ULN, the patient may undergo cardiac evaluation and be considered for treatment
* Patients must not have known hypersensitivity to nivolumab and BMS-986016 or compounds of similar chemical or biologic composition
* Patients must not have a history of severe hypersensitivity reaction to any monoclonal antibody
* Patients must have had prior therapy on PD-1/PD-L1 therapy with progression on therapy or within 6 months of completion of PD-1/PD-L1 inhibitor therapy
* Patients must not have a history of toxic epidermal necrolysis (Stevens-Johnson syndrome)
* Patients must not have received growth factors, including but not limited to granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin, etc. within 2 weeks of study drug administration. Use of such agents while on study is also prohibited. Prior use of growth factors should be documented in the patient's medical history
* Patients must not have a history of any autoimmune disease: inflammatory bowel disease, (including ulcerative colitis and Crohn's disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus (SLE) autoimmune vasculitis (e.g., Wegener's granulomatosis), central nervous system (CNS) or motor neuropathy considered to be of autoimmune origin (e.g., Guillian-Barre syndrome, myasthenia gravis, multiple sclerosis). Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event). Entry of patients with autoimmune diagnoses not listed here must be approved by the protocol chair
* Patients must not be on supplemental home oxygen
* Patients must not have prior treatment with anti-LAG3 inhibitors
* Patients must not have evidence of interstitial lung disease
* Patients with a requirement for steroid treatment or other immunosuppressive treatment: Patients will be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Patients must not not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for at least one week prior to the start of treatment and for the duration of study participation. Patients of childbearing potential must continue to use accepted and effective methods of contraception for 5 months after the last dose of protocol treatment. In addition, patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to registration with a minimum sensitivity of at least 50 IU/L and it must be repeated within 24 hours prior to the first dose of nivolumab and BMS-986016. Patients must also not donate sperm while on study treatment. These supersede the requirements in the EAY131 MASTER protocol eligibility section regarding pregnancy testing and contraception requirements.
* Patients with hepatitis B virus (HBV) or hepatitis C virus (HCV) infection may be eligible provided they have the following:

  * There must be no evidence of clinically significant hepatic injury from hepatitis virus infection
  * For HBV, patients must be on suppressive therapy and have undetectable HBV viral load
  * For HCV, patients must either be on suppressive therapy for HCV or have already completed therapy thought to have eradicated HCV
* Patients must meet one of the following criteria:

  * Patients must have tumor amenable to image guided or direct vision biopsy and be willing and able to undergo a tumor biopsy to obtain tissue for research. Biopsy must not be considered to be more than minimal risk to the patient OR
  * Patient will be undergoing a procedure due to medical necessity prior to start of treatment during which the tissue may be collected OR
  * Formalin-fixed paraffin-embedded tumor tissue block(s) or unstained sectioned slides are available for submission following pre-registration. Criteria for the submission of formalin-fixed paraffin-embedded (FFPE) tissue are:

    * Tissue must have been collected within 6 months prior to pre-registration to step 0
    * Collection of the tissue was after the completion of PD-1/PD-L1 therapy
    * Formalin-fixed paraffin-embedded tumor tissue block(s) must meet the minimum requirements outlined in the Master Protocol.

      * NOTE: If tissue submitted for central LAG-3 testing meets this criteria, additional tissue is not necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. 90% two-sided confidence interval is calculated for ORR. For the purposes of this study, patients should be re-evaluated for response:
  * For treatments given in 21 day (3 week) cycles: every 3 cycles (9 weeks) for the first 33 cycles, and every 4 cycles thereafter (12 weeks)
  * For treatments given in 28 day (4 week) cycles: every 2 cycles (8 weeks) for the first 26 cycles, and every three cycles thereafter (12 weeks)
  * For treatments given in 42 day (6 week) cycles: every 2 cycles (12 weeks)

SECONDARY OUTCOMES:
Overall survival (OS) | From start of treatment on that step until death, or censored at the date of last contact, assessed up to 3 years
  Will be evaluated specifically for each drug (or step). OS will be estimated using the Kaplan-Meier method.
6-month progression free survival (PFS) | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed at 6 months
  Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Progression free survival | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed up to 3 years
  PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer S Azad, Principal Investigator — ECOG-ACRIN Cancer Research Group

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm